CLINICAL TRIAL: NCT03784443
Title: Combined Anti-VEGF Intravitreal Injections With Sustained Steroid Implantation for the Treatment of Diabetic Macular Oedema
Brief Title: Combined Ranibizumab and Iluvien for Diabetic Macular Oedema
Acronym: CASSIE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funder withdrawn funding.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P78912
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Macular Edema; Diabetes
Keywords: Diabetes; Eye; Macular Oedema; Intravitreal Injection; Ranibizumab; Fluocinolone Acetonide
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Fluocinolone Acetonide; Drug Implants; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Double masking randomized control trial with 2 parallel treatment arms: intervention (Iluvien plus Ranibizumab) vs control (Sham plus Ranibizumab)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To maintain double-masking, participants assigned to the control arm will receive sham implantation. This will be performed with an empty Luer Lock Syringe without a needle attached to it, that will not penetrate the eye nor deliver any drug.
  The Iluvien and the sham injection should be performed by the unmasked investigator. The unmasked investigator should not be involved in any patient assessment in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iluvien Arm (Active Comparator): Participants assigned to the Iluvien treatment arm will receive Iluvien 0.19 MG Drug Implant to the study eye under aseptic condition at baseline visit with monthly Ranibizumab Injection [Lucentis] for first three visits followed by monthly Ranibizumab Injection [Lucentis] PRN.
  Interventions: Drug: Iluvien 0.19 MG Drug Implant; Drug: Ranibizumab Injection [Lucentis]
- Control Arm (Sham Comparator): To maintain double-masking, participants assigned to the control arm will receive Sham Intravitreal Injection at the baseline visit with monthly Ranibizumab Injection [Lucentis] for first three visits followed by monthly Ranibizumab Injection [Lucentis] PRN.
  Interventions: Drug: Ranibizumab Injection [Lucentis]; Procedure: Sham Intravitreal Injection

INTERVENTIONS:
Drug: Iluvien 0.19 MG Drug Implant — Fluocinolone Acetonide Sustained Release Intravitreal Implant at Baseline Visit
  Other Names: Fluocinolone Acetonide Implant
  Arms: Iluvien Arm
Drug: Ranibizumab Injection [Lucentis] — Monthly PRN intravitreal injections
  Other Names: Lucentis
Procedure: Sham Intravitreal Injection — Sham injection without penetrating needle and without drug delivery at baseline visit.
  Other Names: Sham Injection with Luer Lock Syringe
  Arms: Control Arm

SUMMARY:
This trial investigated whether adding Iluvien sustained release steroid intravitreal eye implant at the beginning of regular anti-VEGF (anti Vascular Endothelial Growth Factor) intravitreal eye injection treatment for diabetic macular oedema would improve disease stability and reduce the need for regular anti-VEGF intravitreal eye injections over first two years. Diabetic macular oedema, accumulation of microscopic fluid at the back of the eye, is a major cause of poor vision in patients with diabetes.

This is a double mask randomized control multisite trial, to be conducted at 10 NHS hospital eye clinics in England.

DETAILED DESCRIPTION:
This study will recruit 58 participants in a double-masked, multi-centre, sham-controlled clinical trial. Participants will receive Iluvien implantation or sham implantation (masked) with a concomitant intravitreal injection of ranibizumab at baseline with an allocation ratio of 1:1. This is followed by regular monthly clinic review and repeat intravitreal ranibizumab injections to the study eye according to a PRN (pro re nata) treatment protocol.

This trial aims to evaluate whether Iluvien implantation in addition to standard anti-VEGF injection treatment for diabetic macular oedema in pseudophakic eyes will show similar visual acuity outcomes but with an improved reduction in CRT (Central Retinal Thickness) while reducing the average number of intravitreal injections during the first 2 years of treatment, due to the continual micro-dosing of Iluvien therapy.

Participants meeting all the eligibility criteria will be randomized to either Iluvien implant or sham implant procedure with an allocation ratio of 1:1. Participants assigned to either treatment arms will receive intravitreal injection of ranibizumab after Iluvien implantation or sham implantation at the same baseline visit.

To maintain double-masking, participants assigned to the control arm will receive sham implantation. This will be performed with an empty Luer Lock Syringe without a needle attached to it, that will not penetrate the eye nor deliver any drug. Patients assigned to either treatment arm will receive ranibizumab intravitreal injection to the study eye at baseline 30 minutes after the Iluvien or sham implantation. The sham injection should be performed by the unmasked investigator. The unmasked investigator should not be involved in any patient assessment in the study.

Participants will be followed up monthly for 2 years. Participants from both arms will receive compulsory Ranibizumab injection during the first three monthly visit and followed by monthly Ranibizumab as per PRN protocol. The end of study visit should take place at 104 weeks from the baseline visit.

Visual acuity measurement should be performed by trial certified optometrist according to the standard ETDRS (Early Treatment of Diabetic Retinopathy Study) protocol. This is to be conducted in certified examination rooms.

Spectral domain OCT (Optical Coherence Tomography) should be used to assess diabetic macular oedema and optic disc morphology at each visit. The OCT viewer software should be able to provide objective retinal thickness measurement of the central 1mm subfield thickness. Technicians should check for segmentation errors with every OCT scan and make appropriate manual adjustments.

OCT machines and designated technicians at each site will be certified prior to study commencement. Patients must always be assessed using the same OCT model.

7-View Fundus Photography and Fluorescein Angiography (FA) will be performed at the screening visit to confirm the diagnosis of diabetic macular oedema and assess diabetic retinopathy.

Additional FAs may be undertaken during subsequent visits should the investigator believe that there is a clinical need for it. Investigators at each local site are responsible for FA and OCT image interpretation. There will be no centralized image reading centre involved in this study.

IOP (Intraocular Pressure) measurement should be performed with Goldman tonometry either with undilated or dilated pupils.

The primary outcome analysis will be performed to test the differences in the average number of intravitreal injections between the two treatment arms up to month 24. This will be carried out according to an intent to treat principle.

The change of visual acuity from baseline to month 24 will be tested for non-inferiority against the control arm. We will analyze the stability of visual acuity and CRT using AUC (Area Under Curve) Analysis and estimate the average cost of resources utilization for both treatment arms.

Methods of dealing with missing data will follow established techniques, using multiple imputation to impute missing data. If necessary sensitivity analyses will be undertaken to examine the dependence of the results on the method of imputation.

ELIGIBILITY:
Inclusion Criteria:

General

1. Willingness and the ability to provide informed consent.
2. Ability and willingness to undertake all scheduled visits, assessment and treatment.
3. Age 18 years or above.
4. Documented diagnosis of diabetes mellitus (Type I or Type II) as per WHO (World Health Organization) criteria.
5. Current regular use of oral anti-hyperglycaemia or insulin therapy.
6. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year during the study duration of 24 months.

Ocular

1. Macular thickening due to Diabetic Macular Oedema (DMO) involving the centre of fovea as measured by Spectral Domain OCT with CRT of at least 400 microns.
2. DMO confirmed by clinical examination and fundus fluorescein angiography.
3. BCVA between 73 to 25 letters inclusive (Snellen equivalent to 6/12 to 6/96) as measured using ETDRS protocol at 4 meters.
4. Pseudophakia in the study eye.
5. Adequate ocular media clarity and pupillary dilatation allowing for posterior segment examination and OCT scanning.

Exclusion Criteria:

General

1. Cerebral vascular accident, transient ischaemic attack or myocardial infarction within 3 months prior to day 1 (baseline).
2. Pregnancy or breastfeeding, or intention to become pregnant during the study.
3. Participation in an investigational trial involving treatment with any drug or devices within 3 months prior to day 1 (baseline) and must not be enrolled in another investigational trial during their participation in this trial.
4. Systemic anti-VEGF-base therapies within 3 months prior to day 1 (baseline).

Ocular

1. History of prior intravitreal anti-VEGF therapy or steroid implant in the study eye.
2. History of proliferative diabetic retinopathy.
3. History of rubeosis or current rubeosis.
4. History of neovascularization, tractional retinal detachment, retinal vein occlusion, or significant pre-retinal fibrosis distorting the macular architecture.
5. History of retinal detachment or macular hole stage 3 or above.
6. History of vitreoretinal surgery.
7. Aphakia.
8. History of glaucoma or uncontrolled ocular hypertension.
9. Active or suspected ocular or periocular infection or inflammation, including viral diseases of the cornea, conjunctiva and retina, such as active epithelial herpes simplex keratitis (dendritic keratitis), varicella, mycobacterial infections, and fungal diseases.
10. Panretinal Photocoagulation (PRP) laser treatment within 3 months prior to day 1.
11. Macular laser (focal or grid) within 3 months prior to day 1.
12. YAG (yttrium aluminium garnet) laser capsulotomy laser within 3 months prior to day 1.
13. Any periocular steroid treatment within 6 months prior to day 1.
14. Cataract operation within 3 months prior to day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Lucentis Injections received in the study eye | 24 months
  The total number of Lucentis injections needed over 24 months following the intravitreal injection PRN protocol

SECONDARY OUTCOMES:
Change in visual acuity | Month 24
  Change in ETDRS (Early Treatment of Diabetic Retinopathy Study) best corrected visual acuity from baseline to month 24
Maintaining at least 20/40 vision | Month 24
  Percentage of patients that achieve or maintain 20/40 vision
Proportion of participants with vision loss | Month 24
  Proportion of participants losing 5, 10, 15 ETDRS letters or more
Proportion of participants with visual gain | Month 24
  Proportion of participants gaining at least 5, 10, 15 ETDRS letters or more
Stability of vision | Over 24 months
  Stability of visual acuity over 24 months using Area Under Curve Analysis (AUC)
Central retinal thickness | Month 24
  Central retinal thickness (CRT) change as measured by Spectral Domain OCT
CRT stability | Over 24 months
  Stability of CRT over 24 months using AUC analysis
Retinal thickness variability | Over 24 months
  The difference between min and max retinal thickness
Change in Diabetic Retinopathy Severity | Between baseline and month 24
  Measured using the ETDRS DRSS (Diabetic Retinopathy Severity Score)
Number of focal laser treatments | Over 24 months
  Number of focal laser treatments

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cheong-Leen, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antonetti DA, Klein R, Gardner TW. Diabetic retinopathy. N Engl J Med. 2012 Mar 29;366(13):1227-39. doi: 10.1056/NEJMra1005073. No abstract available. PMID 22455417
- [Background] Bunce C, Wormald R. Causes of blind certifications in England and Wales: April 1999-March 2000. Eye (Lond). 2008 Jul;22(7):905-11. doi: 10.1038/sj.eye.6702767. Epub 2007 Mar 2. PMID 17332762
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648
- [Background] Yau JW, Rogers SL, Kawasaki R, Lamoureux EL, Kowalski JW, Bek T, Chen SJ, Dekker JM, Fletcher A, Grauslund J, Haffner S, Hamman RF, Ikram MK, Kayama T, Klein BE, Klein R, Krishnaiah S, Mayurasakorn K, O'Hare JP, Orchard TJ, Porta M, Rema M, Roy MS, Sharma T, Shaw J, Taylor H, Tielsch JM, Varma R, Wang JJ, Wang N, West S, Xu L, Yasuda M, Zhang X, Mitchell P, Wong TY; Meta-Analysis for Eye Disease (META-EYE) Study Group. Global prevalence and major risk factors of diabetic retinopathy. Diabetes Care. 2012 Mar;35(3):556-64. doi: 10.2337/dc11-1909. Epub 2012 Feb 1. PMID 22301125
- [Background] Virgili G, Parravano M, Menchini F, Evans JR. Anti-vascular endothelial growth factor for diabetic macular oedema. Cochrane Database Syst Rev. 2014 Oct 24;(10):CD007419. doi: 10.1002/14651858.CD007419.pub4. PMID 25342124
- [Background] Grover D, Li TJ, Chong CC. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD005656. doi: 10.1002/14651858.CD005656.pub2. PMID 18254088
- [Background] Goni FJ, Stalmans I, Denis P, Nordmann JP, Taylor S, Diestelhorst M, Figueiredo AR, Garway-Heath DF. Elevated Intraocular Pressure After Intravitreal Steroid Injection in Diabetic Macular Edema: Monitoring and Management. Ophthalmol Ther. 2016 Jun;5(1):47-61. doi: 10.1007/s40123-016-0052-8. Epub 2016 May 10. PMID 27164896
- [Background] Parrish RK 2nd, Campochiaro PA, Pearson PA, Green K, Traverso CE; FAME Study Group. Characterization of Intraocular Pressure Increases and Management Strategies Following Treatment With Fluocinolone Acetonide Intravitreal Implants in the FAME Trials. Ophthalmic Surg Lasers Imaging Retina. 2016 May 1;47(5):426-35. doi: 10.3928/23258160-20160419-05. PMID 27183546
- [Background] Funatsu H, Yamashita H, Ikeda T, Mimura T, Eguchi S, Hori S. Vitreous levels of interleukin-6 and vascular endothelial growth factor are related to diabetic macular edema. Ophthalmology. 2003 Sep;110(9):1690-6. doi: 10.1016/S0161-6420(03)00568-2. PMID 13129863
- [Background] Funatsu H, Yamashita H, Sakata K, Noma H, Mimura T, Suzuki M, Eguchi S, Hori S. Vitreous levels of vascular endothelial growth factor and intercellular adhesion molecule 1 are related to diabetic macular edema. Ophthalmology. 2005 May;112(5):806-16. doi: 10.1016/j.ophtha.2004.11.045. PMID 15878060
- [Background] Aiello LP. Angiogenic pathways in diabetic retinopathy. N Engl J Med. 2005 Aug 25;353(8):839-41. doi: 10.1056/NEJMe058142. No abstract available. PMID 16120866
- [Background] Wang K, Wang Y, Gao L, Li X, Li M, Guo J. Dexamethasone inhibits leukocyte accumulation and vascular permeability in retina of streptozotocin-induced diabetic rats via reducing vascular endothelial growth factor and intercellular adhesion molecule-1 expression. Biol Pharm Bull. 2008 Aug;31(8):1541-6. doi: 10.1248/bpb.31.1541. PMID 18670086
- [Background] Minassian DC, Owens DR, Reidy A. Prevalence of diabetic macular oedema and related health and social care resource use in England. Br J Ophthalmol. 2012 Mar;96(3):345-9. doi: 10.1136/bjo.2011.204040. Epub 2011 May 20. PMID 21602478
- [Background] Arevalo JF, Lasave AF, Wu L, Acon D, Farah ME, Gallego-Pinazo R, Alezzandrini AA, Fortuna V, Quiroz-Mercado H, Salcedo-Villanueva G, Maia M, Serrano M, Rojas S; Pan-American Collaborative Retina Study Group (PACORES). Intravitreal bevacizumab for diabetic macular oedema: 5-year results of the Pan-American Collaborative Retina Study group. Br J Ophthalmol. 2016 Dec;100(12):1605-1610. doi: 10.1136/bjophthalmol-2015-307950. Epub 2016 Feb 24. PMID 26912377
- [Background] Wells JA, Glassman AR, Ayala AR, Jampol LM, Bressler NM, Bressler SB, Brucker AJ, Ferris FL, Hampton GR, Jhaveri C, Melia M, Beck RW; Diabetic Retinopathy Clinical Research Network. Aflibercept, Bevacizumab, or Ranibizumab for Diabetic Macular Edema: Two-Year Results from a Comparative Effectiveness Randomized Clinical Trial. Ophthalmology. 2016 Jun;123(6):1351-9. doi: 10.1016/j.ophtha.2016.02.022. Epub 2016 Feb 27. PMID 26935357
- [Background] Mehta H, Gillies M, Fraser-Bell S. Perspective on the role of Ozurdex (dexamethasone intravitreal implant) in the management of diabetic macular oedema. Ther Adv Chronic Dis. 2015 Sep;6(5):234-45. doi: 10.1177/2040622315590319. PMID 26336592
- [Background] Hernandez-Bel L, Cervera-Taulet E, Navarro-Palop C, Castro-Navarro V, Chiarri-Toumit C, Montero-Hernandez J. Sequential Dexamethasone and Aflibercept Treatment in Patients with Diabetic Macular Edema: Structural and Functional Outcomes at 52 Weeks. Ophthalmologica. 2019;241(2):98-104. doi: 10.1159/000489345. Epub 2018 Jul 11. PMID 29996128
- [Background] Campochiaro PA, Brown DM, Pearson A, Chen S, Boyer D, Ruiz-Moreno J, Garretson B, Gupta A, Hariprasad SM, Bailey C, Reichel E, Soubrane G, Kapik B, Billman K, Kane FE, Green K; FAME Study Group. Sustained delivery fluocinolone acetonide vitreous inserts provide benefit for at least 3 years in patients with diabetic macular edema. Ophthalmology. 2012 Oct;119(10):2125-32. doi: 10.1016/j.ophtha.2012.04.030. Epub 2012 Jun 21. PMID 22727177
- [Background] Cunha-Vaz J, Ashton P, Iezzi R, Campochiaro P, Dugel PU, Holz FG, Weber M, Danis RP, Kuppermann BD, Bailey C, Billman K, Kapik B, Kane F, Green K; FAME Study Group. Sustained delivery fluocinolone acetonide vitreous implants: long-term benefit in patients with chronic diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1892-903. doi: 10.1016/j.ophtha.2014.04.019. Epub 2014 Jun 14. PMID 24935282
- [Background] Shimura M, Yasuda K, Minezaki T, Noma H. Reduction in the frequency of intravitreal bevacizumab administrations achieved by posterior subtenon injection of triamcinolone acetonide in patients with diffuse diabetic macular edema. Jpn J Ophthalmol. 2016 Sep;60(5):401-7. doi: 10.1007/s10384-016-0458-9. Epub 2016 Jun 15. PMID 27306783
- [Background] Prunte C, Fajnkuchen F, Mahmood S, Ricci F, Hatz K, Studnicka J, Bezlyak V, Parikh S, Stubbings WJ, Wenzel A, Figueira J; RETAIN Study Group. Ranibizumab 0.5 mg treat-and-extend regimen for diabetic macular oedema: the RETAIN study. Br J Ophthalmol. 2016 Jun;100(6):787-95. doi: 10.1136/bjophthalmol-2015-307249. Epub 2015 Oct 9. PMID 26453639